CLINICAL TRIAL: NCT07014371
Title: Alternative vs. Once-Daily Oral Iron Supplementation in Iron Deficiency Anemia (IDA): A Multicenter, Randomized, Open-Label, Non-Inferiority Trial
Brief Title: Alternative vs. Once-Daily Oral Iron Supplementation in Iron Deficiency Anemia (IDA)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hemato-001
Record Dates: First submitted 2025-06-01; First posted 2025-06-11 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Iron Deficiency Anemia Treatment
Keywords: Iron deficiency anemia; Ferrous fumarate; Alternate day dosing; Hemoglobin
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferrous fumarate; Tablets; Iron-Dextran Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Once-Daily Dosing Group (Active Comparator): Participants will receive ferrous fumarate 200 mg, taken orally once daily for 8 weeks. This arm represents the standard dosing regimen for treating iron deficiency anemia (IDA). Participants will be monitored at baseline, Week 4, and Week 8 for blood counts, iron parameters, and adverse effects. Medication adherence will be assessed using pill counts.
  Interventions: Drug: Ferrous Fumarate Oral Tablet
- Alternate-Day Dosing Group (Experimental): Participants will receive ferrous fumarate 400 mg (two 200 mg tablets), taken orally on alternate days for 8 weeks. This dosing strategy is being evaluated for improved iron absorption and fewer gastrointestinal side effects compared to daily dosing. Participants will be monitored at baseline, Week 4, and Week 8 for blood counts, iron parameters, and adverse effects. Medication adherence will be assessed using pill counts.
  Interventions: Drug: Ferrous Fumarate Oral Tablet

INTERVENTIONS:
Drug: Ferrous Fumarate Oral Tablet — Ferrous fumarate oral tablet 200 mg is an iron supplement used for the treatment of iron deficiency anemia (IDA). In this study, it is administered as either one tablet daily (OD group) or two tablets on alternate days (AD group), with a treatment duration of 8 weeks. The goal is to compare the efficacy and tolerability of alternate-day dosing versus standard once-daily dosing.
  Other Names: Ferrous Fumarate 200 mg tablet; Oral iron supplement

SUMMARY:
The goal of this clinical trial is to compare the effectiveness and tolerability of two different oral iron regimens in adults with iron deficiency anemia (IDA). The main questions it aims to answer are:

Is alternate-day oral iron supplementation as effective as once-daily dosing in improving hemoglobin levels?

What are the side effects associated with each dosing regimen?

Researchers will compare once-daily vs. alternate-day oral ferrous fumarate to evaluate whether alternate-day dosing is non-inferior in terms of hematologic response, with fewer adverse effects.

Participants will:

Be randomly assigned to take ferrous fumarate 200 mg once daily or 400 mg on alternate days for 8 weeks

Undergo blood tests and clinical assessments at baseline, Week 4, and Week 8

Report any side effects and bring remaining pills to evaluate medication adherence

This is a multicenter, randomized, open-label, non-inferiority trial conducted in adults aged 20 years or older with IDA.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥20 years diagnosed with iron deficiency anemia, defined as: hemoglobin (Hb) <13 g/dL in males or <12 g/dL in females, and ferritin <50 ng/mL or transferrin saturation (TSAT) <20%.
* No iron supplementation within the past 3 months.

Exclusion Criteria:

* Hemodynamic instability (e.g., acute bleeding or hypotension).
* Severe heart failure (New York Heart Association [NYHA] Class III-IV) or other active cardiac diseases.
* Active malignancy or history of cancer within the past 3 years (except non-melanoma skin cancer).
* Pregnancy or breastfeeding.
* Chronic liver disease including cirrhosis (Child-Pugh class B or C).
* Chronic kidney disease (estimated glomerular filtration rate [eGFR] <60 mL/min/1.73 m²).
* Clinically significant thalassemia or hemoglobinopathies.
* Ongoing infection or chronic inflammatory diseases (e.g., rheumatoid arthritis, inflammatory bowel disease).
* Malabsorption disorders (e.g., history of bariatric surgery).
* Red blood cell transfusion within the past 3 months.

Withdrawal Criteria

* Withdrawal of informed consent.
* Severe adverse events requiring permanent discontinuation of study medication.
* Investigator's judgment that continued participation poses a safety risk.
* Non-adherence to study medication (compliance < 75%).

Treatment Failure

- Increase in hemoglobin level of < 1 g/dL at Week 4 or Week 8 compared with baseline.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin Level at Week 8 After Oral Iron Supplementation | 8 weeks
  Hemoglobin concentration (g/dL) measured at Week 8 following oral ferrous fumarate supplementation. Participants are stratified by sex and baseline Hb level. Comparison between once-daily and alternate-day dosing groups will be analyzed using a linear mixed-effects model.

SECONDARY OUTCOMES:
Change in Reticulocyte Count at Weeks 4 and 8 | 4 and 8 weeks
  Mean change in reticulocyte count (%) from baseline to Week 4 and Week 8.
Change in Serum Ferritin at Weeks 4 and 8 | 4 and 8 weeks
  Mean change in serum ferritin concentration (ng/mL) from baseline to Week 4 and Week 8.
Adverse Effects of Ferrous Fumarate | During the 8-week treatment period
  Incidence and type of adverse effects experienced by participants during treatment with ferrous fumarate oral tablets.

CONTACTS AND LOCATIONS:
Locations (1):
- Phramongkutklao Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to institutional policy and privacy concerns. Only aggregate data may be shared upon reasonable request.